CLINICAL TRIAL: NCT05974501
Title: Pre vs. Postoperative Adductor Canal Block for Total Knee Arthroplasty: Prospective Randomized Trial
Brief Title: Pre vs Post Block in Total Knee Arthroplasty (TKA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Victor Hugo Hernandez, Professor of Clinical, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 20230147
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Results first posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: Knee Osteoarthritis; Arthroplasty Complications; Postoperative Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain, Postoperative | interventions — Dexamethasone; Acetaminophen; Pregabalin; Celecoxib; Meloxicam; Oxycodone; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preoperative Adductor Canal Block Group (Active Comparator): Participants in this group will receive the standard of care treatment for pain management for TKA including a preoperative adductor canal block. Participants will be in this group for up to 24 hours after surgery.
  Interventions: Drug: Dexamethasone; Drug: Acetaminophen; Drug: Lyrica; Drug: Celebrex; Drug: Meloxicam; Drug: Oxycodone; Drug: Ropivacaine
- Postoperative Adductor Canal Block Group (Experimental): Participants in this group will receive the standard of care treatment for pain management after TKA, however, the adductor canal block will be placed postoperatively. Participants will be in this group for up to 24 hours
  Interventions: Drug: Dexamethasone; Drug: Acetaminophen; Drug: Lyrica; Drug: Celebrex; Drug: Meloxicam; Drug: Oxycodone; Drug: Ropivacaine

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 10mg administered via IV once postoperatively within 24 hours for pain and swelling
Drug: Acetaminophen — 1,000mg administered via tablet every 8 hours for pain during the first 1-2 weeks postoperatively
Drug: Lyrica — Administered via tablet 75mg nightly for pain during the first 1-2 weeks postoperatively
Drug: Celebrex — 200mg administered via tablet twice a day for pain and swelling during the first 1-2 weeks postoperatively
Drug: Meloxicam — 30mg administered via IV once postoperatively within 24 hours for pain and swelling
Drug: Oxycodone — 5mg administered via tablet every 4 hours as needed for pain during the first 1-2 weeks postoperatively
Drug: Ropivacaine — 20 milliliters Ropivacaine 0.2% administered via injection perioperatively.
  Other Names: Adductor Canal Block

SUMMARY:
The purpose of this project is to determine if a change in patient reported pain, nausea and vomiting after total knee arthroplasty can be observed with the substitution of a post operative adductor canal block for a preoperative adductor canal block in the current established peri-operative pain protocol and if these changes lead to a decrease in opioid consumption (in morphine equivalents).

ELIGIBILITY:
Inclusion Criteria:

1- Patients 18 or older 2 - Patients undergoing primary total knee replacement at the University of Miami Hospital 3 - Patients that have capacity to provide medical consent

Exclusion Criteria:

1. All patients under the age of 18
2. Prisoners, uncontrolled diabetics, increased risk of bleeding, pregnant women, women planning on becoming pregnant in the next year, and women who think they might be pregnant.
3. Patients with prior surgery or history of infection on the joint of interest.
4. Patients on steroid preoperatively.
5. Inability to provide medical consent.
6. Patients with a history of significant unmitigated pain in parts of their body not including the knee the procedure is to be performed or a history of pain catastrophizing (the tendency to magnify the threat value of the pain stimulus and to feel helpless in the context of pain, and by a relative inability to inhibit pain-related thoughts in anticipation of, during or following a painful event) regarding pain anywhere in the body.
7. Any condition that, in the opinion of the investigator, would compromise the well-being of the patient or the study or prevent the patient from meeting or performing study requirements will exclude the participant.
8. Allergy to local anesthetic or any medication used in the standard protocol for joint replacement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-09-29 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor H. Hernandez, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Preoperative Adductor Canal Block Group | Postoperative Adductor Canal Block Group
Started | 46 | 38
Completed | 46 | 37
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: The number of individual patients in the respective group
Groups:
- Total: Total of all reporting groups
Arm/Group | Preoperative Adductor Canal Block Group | Postoperative Adductor Canal Block Group | Total
Number analyzed (Participants) | 46 | 38 | 84
Age, Continuous [Median (Standard Deviation); unit: years] | 65 (9.12) | 65 (9.75) | 65 (9.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 26 | 57
  Male | 15 | 12 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (BMI) [Median (Standard Deviation); unit: kg/m^2] | 30.50 (4.73) | 30.90 (4.18) | 30.80 (4.51)

OUTCOME MEASURES:

1. Primary Outcome: Pain Status as Measured by Numeric Pain Scale
Description: Scale with numeric scores ranging from 0 (least) to 10 (most) pain
Time Frame: 2 hours postoperatively
Population: Patients who completed the study in one of the two groups
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Preoperative Adductor Canal Block Group | Postoperative Adductor Canal Block Group
Number analyzed (Participants) | 46 | 37
score on a scale | 2 [1.00 to 6.00] | 4.00 [1.00 to 5.00]

2. Primary Outcome: Pain Status as Measured by Numeric Pain Scale
Description: Scale with numeric scores ranging from 0 (least) to 10 (most) pain
Time Frame: 24 hours postoperatively
Population: Patients who completed the study in one of the two groups
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Preoperative Adductor Canal Block Group | Postoperative Adductor Canal Block Group
Number analyzed (Participants) | 46 | 37
score on a scale | 6.00 [4.00 to 7.00] | 6.00 [5.00 to 8.00]

3. Secondary Outcome: Patients Reporting Nausea
Description: Count of the number of patients reporting nausea
Time Frame: 2 hours postoperatively
Population: Patients who completed the study in one of the two groups
Measure: Count of Participants; unit: Participants
Arm/Group | Preoperative Adductor Canal Block Group | Postoperative Adductor Canal Block Group
Number analyzed (Participants) | 46 | 37
Participants | 7 | 4

4. Secondary Outcome: Episodes of Nausea
Description: Count of the number of episodes of nausea per patient
Time Frame: 2 hours postoperatively
Population: Patients who completed the study in one of the two groups
Measure: Median (95% Confidence Interval); unit: number of episodes per patient
Arm/Group | Preoperative Adductor Canal Block Group | Postoperative Adductor Canal Block Group
Number analyzed (Participants) | 46 | 37
number of episodes per patient | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

5. Secondary Outcome: Patients Reporting Nausea
Description: Count of the number of patients reporting nausea
Time Frame: 24 hours postoperatively
Population: Patients who completed the study in one of the two groups
Measure: Count of Participants; unit: Participants
Arm/Group | Preoperative Adductor Canal Block Group | Postoperative Adductor Canal Block Group
Number analyzed (Participants) | 46 | 37
Participants | 8 | 5

6. Secondary Outcome: Episodes of Nausea
Description: Count of the number of episodes of nausea per patient
Time Frame: 24 hours postoperatively
Population: Patients who completed the study in one of the two groups
Measure: Median (95% Confidence Interval); unit: number of episodes per patient
Arm/Group | Preoperative Adductor Canal Block Group | Postoperative Adductor Canal Block Group
Number analyzed (Participants) | 46 | 37
number of episodes per patient | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

7. Secondary Outcome: Patients Reporting Vomiting
Description: Count of the number of patients reporting vomiting
Time Frame: 2 hours postoperatively
Population: Patients who completed the study in one of the two groups
Measure: Count of Participants; unit: Participants
Arm/Group | Preoperative Adductor Canal Block Group | Postoperative Adductor Canal Block Group
Number analyzed (Participants) | 46 | 37
Participants | 1 | 1

8. Secondary Outcome: Episodes of Vomiting
Description: Count of the number of episodes of vomiting per patient
Time Frame: 2 hours postoperatively
Population: Patients who completed the study in one of the two groups
Measure: Median (95% Confidence Interval); unit: number of episodes per patient
Arm/Group | Preoperative Adductor Canal Block Group | Postoperative Adductor Canal Block Group
Number analyzed (Participants) | 46 | 37
number of episodes per patient | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

9. Secondary Outcome: Patients Reporting Vomiting
Description: Count of the number of patients reporting vomiting
Time Frame: 24 hours postoperatively
Population: Patients who completed the study in one of the two groups
Measure: Count of Participants; unit: Participants
Arm/Group | Preoperative Adductor Canal Block Group | Postoperative Adductor Canal Block Group
Number analyzed (Participants) | 46 | 37
Participants | 3 | 2

10. Secondary Outcome: Episodes of Vomiting
Description: Count of the number of episodes of vomiting per patient
Time Frame: 24 hours postoperatively
Population: Patients who completed the study in one of the two groups
Measure: Median (95% Confidence Interval); unit: number of episodes per patient
Arm/Group | Preoperative Adductor Canal Block Group | Postoperative Adductor Canal Block Group
Number analyzed (Participants) | 46 | 37
number of episodes per patient | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

11. Secondary Outcome: Total Opioid Consumption
Description: Measure of the amount of morphine milliequivalents consumed by the patient
Time Frame: 2 hours postoperatively
Population: Patients who completed the study in one of the two groups
Measure: Median (95% Confidence Interval); unit: milligram morphine equivalents
Arm/Group | Preoperative Adductor Canal Block Group | Postoperative Adductor Canal Block Group
Number analyzed (Participants) | 46 | 37
milligram morphine equivalents | 19.50 [8.00 to 30.00] | 30.00 [15.00 to 32.00]

12. Secondary Outcome: Total Opioid Consumption
Description: Measure of the amount of morphine milliequivalents consumed by the patient
Time Frame: 24 hours postoperatively
Population: Patients who completed the study in one of the two groups
Measure: Median (95% Confidence Interval); unit: milligram morphine equivalents
Arm/Group | Preoperative Adductor Canal Block Group | Postoperative Adductor Canal Block Group
Number analyzed (Participants) | 46 | 37
milligram morphine equivalents | 45.00 [30.00 to 56.00] | 36.00 [30.00 to 56.00]

13. Secondary Outcome: Nights Hospitalized
Description: Number of nights hospitalized
Time Frame: Up to 14 nights postoperatively
Population: Patients who completed the study in one of the two groups
Measure: Median (95% Confidence Interval); unit: nights
Arm/Group | Preoperative Adductor Canal Block Group | Postoperative Adductor Canal Block Group
Number analyzed (Participants) | 46 | 37
nights | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]

14. Secondary Outcome: Hours Hospitalized
Description: Number of hours hospitalized
Time Frame: Up to 336 hours postoperatively
Population: Patients who completed the study in one of the two groups
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Preoperative Adductor Canal Block Group | Postoperative Adductor Canal Block Group
Number analyzed (Participants) | 46 | 37
hours | 23.66 [21.92 to 25.48] | 25.92 [23.60 to 27.07]

15. Secondary Outcome: Discharges by Midnight POD0
Description: The number of patients discharged home by midnight on postoperative day zero
Time Frame: Up to 24 hours postoperatively
Population: Patients who completed the study in one of the two groups
Measure: Count of Participants; unit: Participants
Arm/Group | Preoperative Adductor Canal Block Group | Postoperative Adductor Canal Block Group
Number analyzed (Participants) | 46 | 37
Participants | 3 | 4

16. Secondary Outcome: Discharges by Midnight on POD1
Description: The number of patients discharged home by midnight postoperative day one
Time Frame: Up to 48 hours postoperatively
Population: Patients who completed the study in one of the two groups
Measure: Count of Participants; unit: Participants
Arm/Group | Preoperative Adductor Canal Block Group | Postoperative Adductor Canal Block Group
Number analyzed (Participants) | 46 | 37
Participants | 40 | 29

ADVERSE EVENTS:
Time Frame: 24 hours postoperatively
Arm/Group | Preoperative Adductor Canal Block Group | Postoperative Adductor Canal Block Group
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/38
Other Adverse Events (participants affected / at risk) | 0/46 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT05974501/Prot_SAP_000.pdf